CLINICAL TRIAL: NCT05493592
Title: Interest of a Diet Rich in Cajanus Cajan (Pigeon Pea) Associated With a Standardized Exercise Protocol on NLRP3 Inflammasome Expression and Weight Loss in Adult Patients With Severe Obesity.
Brief Title: Pigeon Peas (Cajanus Cajan) : a Natural Anti-inflammatory Facilitating Weight Loss in Obese Patients Returning to Sport?
Acronym: OBESICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: GIRCI SOHO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19_RIPH2-29
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Severe Obesity
Keywords: Severe obesity; Cajanus cajan (pigeon pea); Physical exercise; NLRP3 inflammasome; French caribbean population
MeSH Terms: conditions — Obesity, Morbid; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prescription of a standardized 24-week physical activity protocol alone or accompanied by the consumption of 100 grams of pigeon peas (Cajanus cajan) per meal three times a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized physical activity protocol (EXA control group) (No Intervention): Physical activity protocol for 24 weeks. Protocol of dietetics and food hygiene for 24 weeks.
- Standardized physical activity protocol associated with the consumption of Cajanus cajan (EXACAJAN) (Experimental): The EXACAJAN protocol will be continued for 24 weeks. It will combine 3 times a week with 100 grams of pigeon peas in the diet. Protocol of dietetics and food hygiene for 24 weeks.
  Interventions: Biological: Standardized physical activity protocol associated with the consumption of Cajanus cajan (EXACAJAN)

INTERVENTIONS:
Biological: Standardized physical activity protocol associated with the consumption of Cajanus cajan (EXACAJAN) — Supervised re-training by an Adapted Physical Activity (APA) professional combined 100 g of pigeon peas 3 times a week
  Physical activity protocol is standardized. It's the same than in the control arm.
  The preparation of pigeon peas and their consumption will be standardized in terms of species cultivated, geographical origin and culinary preparation.
  A follow-up of the food intakes standardized plus follow-up logbook, recording the weekly pigeon pea intake, will also be filled out by the participant. The addition of 100 grams of pigeon peas to the diet corresponds to an intake of about 980 mg of polyphenols, 360 mg of carotenoids and 570 mg of vitamin C (24). Thus, the patient's diet will be fortified with approximately 420 mg of polyphenols per day. This level of polyphenol supplementation is known to have beneficial effects on human health.
  Arms: Standardized physical activity protocol associated with the consumption of Cajanus cajan (EXACAJAN)

SUMMARY:
Adult obesity is due to an excess of body fat. This corresponds to all the fat in the body (or adipose tissue). It is opposed to the lean mass which corresponds to the weight of muscles, organs and viscera. It is defined from the body mass index (or BMI). BMI is calculated by dividing a person's weight by their height squared.

According to these criteria, the prevalence of obesity has reached 17% of the entire adult population in mainland France (ESTENBAN 2015 study). The prevalence figures for obesity in the French overseas departments are higher than in mainland France. The latest epidemiological data available in Martinique and Guadeloupe (KANNARI 2015 study) show that approximately 60% of the adult population is overweight and 25% of the adult population is obese.

Obesity is considered a chronic disease that increases the risk of cardiovascular and metabolic complications all the more when patients have a BMI ≥ 35 kg/m2, defining severe obesity. When BMI is equal to or exceeds 40 kg/m2, obesity is said to be "morbid" and the risk of cardiovascular complications increases by about 100% to 400% depending on the type of complications. The risk of mortality increases by 50 to 100% compared to the normal weight population.

Obesity and inflammation Adipose tissue accumulates around the abdominal viscera after the fat storage capacity of the subcutaneous territories has been reached. The accumulation of visceral fat is accompanied by a low-grade inflammatory response that is responsible for the secretion of lipid derivatives and mediators toxic to the cardiovascular system and insulin sensitivity. The inflammatory response is characterized by the expression of numerous pro-inflammatory molecules synthesized by adipocytes and immunocompetent single-macrophage cells infiltrating the vascular stroma of adipose tissue. In addition, hyperglycemia and excess lipid intermediates cause the assembly of inflammasomes in the cytosol. Among them, the NLRP3 inflammasome involved in multiple human inflammatory pathologies.

Inflammation opposes weight loss, hence the need to reduce the inflammatory response to facilitate weight loss in obese people.

Pigeon pea, known for its anti-inflammatory properties, is a legume found in Creole gardens and traditionally eaten at Christmas.

The OBESICA study aims at studying the interest of consuming pigeon pea associated with regular physical activity on the inflammatory state of the body and weight loss in obese patients.

DETAILED DESCRIPTION:
Obesity is a generic term for excess body fat. In adults, the World Health Organization (WHO) defines overweight and obesity by a body mass index (BMI) ≥ 25 kg/m2 and 30 kg/m2, respectively. According to these criteria, the prevalence of obesity has reached 17% of the entire adult population in France (ESTENBAN 2015 study). Obesity prevalence figures in the French overseas departments are higher than in France : 60% of the adult population in Martinique and Guadeloupe is overweight and 25% of the adult population is obese (KANNARI 2015 study).

Obesity increases the risk of cardiovascular and metabolic complications even more when patients have a BMI ≥ of 35 kg/m2, defining severe obesity. When the BMI is equal to or greater than 40 kg/m2, obesity is said to be "morbid" and the risk of cardiovascular complications increases by between 100% and 400% depending on the type of complications. The risk of mortality increases in the order of 50 to 100% compared to the normal weight population. However, some individuals do not present cardio-metabolic abnormalities despite a significant excess of fat.

Several studies show that cardiovascular and metabolic complications are indeed linked to the accumulation of abdominal visceral fat.

An abdominal girth ≥ 94 cm in men and ≥ 80 cm in women defines abdominal obesity and predicts a high risk of cardiovascular complications. While in France, abdominal obesity affects about 40% of adults, it affects 47% of men and up to 70% of women in overseas territories.

The accumulation of visceral fat is accompanied by a low-grade inflammatory response that is responsible for the secretion of lipid derivatives and mediators that are toxic to the cardiovascular system and insulin sensitivity.

The inflammatory response is characterized by the expression of numerous pro-inflammatory molecules synthesized in particular by adipocytes. In addition to the activation of nuclear transcription factors such as NFκB and AP-1, metabolic danger signals such as hyperglycemia and excess lipid intermediates induce the assembly of multi-protein platforms in the cytosol called inflammasomes including the NLRP3 inflammasome.

Activation of the NLRP3 inflammasome activates caspase-1 which its proteolytic activity is responsible for the release of the cytokines IL-1β and IL-18 into tissue and circulating blood.

Strategies that decrease the inflammatory state and the volume of intra-abdominal fat are a therapeutic goal to limit the occurrence of cardiovascular complications and insulin resistance in the obese.

In this context, it is suggested that reducing the inflammatory response could improve weight loss in obese people. Regular physical activity and a healthy diet have clearly demonstrated anti-inflammatory effects and are effective in weight loss in obese patients.

Several epidemiological and clinical studies highlight the potential "health" effects of molecules with anti-inflammatory and antioxidant properties contained in fruits and vegetables, called phyto-micronutrients. In obese patients, phyto-micronutrients such as certain polyphenols of the flavonoid class are beneficial on plasma markers of inflammation, insulin resistance, lipid profile and weight loss. Among legume seeds, Cajanus cajan or pigeon pea represents an interesting variety because of its high content of non-thermosensitive flavonoids of the isoflavone type (genistein and daidzein). In the French Overseas Departments (DOMs).

We hypothesize that the resumption of adapted physical activity and the reintroduction of polyphenol-rich tropical legume seeds in the diet could bring a benefit in the management of severe obesity in overseas territories by reducing the activation of inflammation mediated by the NLRP3 inflammasome and facilitating the reduction of abdominal visceral fat and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI ≥ 35 kg/m² (severely obese)
* Ability, at the time of inclusion, to follow a personalized physical activity program for 24 weeks.
* Have agreed to follow-up for up to 36 weeks
* Be affiliated to a social security system
* Be able to freely give informed consent (oral)

Exclusion Criteria:

* Pregnant woman
* Have a history of type 1 diabetes
* Weight >150 kg (criterion related to the capacity of the exercise bikes used in the study)
* History of renal disease [glomerular filtration < 30 mL/min], cardiovascular history of myocardial ischemia (ECG signs), uncontrolled hypertension [at rest; systolic blood pressure > 140 mm Hg and diastolic blood pressure > 90 mm Hg], heart failure, cardiac valvulopathy, peripheral arterial disease or arteritis, and stroke.
* Have an auto-inflammatory or autoimmune pathology known to modify the expression of NLRP3 (cryopyrinopathies, Crohn's disease, gouty arthritis, chondrocalcinosis, arthritic diseases, type 1 diabetes, Biermer's disease, Basedow's disease, rheumatoid arthritis, systemic lupus erythematosus, sclerodermias, non-alcoholic liver steatosis, multiple sclerosis, Alzheimer's and Parkinson's diseases)
* Have a history of recent (<6 months) infectious disease of viral, parasitic, fungal or bacterial origin known to modify the expression of NLRP3
* Taking medication that may affect weight gain (systemic corticosteroids, psychotropic drugs, migraine medications, beta-blockers, chemotherapy, and antibiotics)
* Have completed a personalized physical activity program in the 12 weeks prior to inclusion,
* Have bariatric surgery scheduled within 6 months of inclusion,
* Have a known intolerance to legume seeds
* Have an unbalanced low-calorie diet
* Have consumed dietary supplements containing polyphenols of the flavonoid class (green tea catechins and isoflavones from soy and legume seeds in the 3 months prior to inclusion).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 124 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of NLRP3 expression | Randomization, 6 and 9 months +/- 8 days post randomisation
  Basal level variation in mRNA expression of the NLRP3 gene (coding for the NLRP3 protein subunit of the NLRP3 inflammasome), in monocytes isolated from peripheral blood. This variation will be measured by RT-qPCR (Quantitative reverse transcription PCR) and will be expressed in DNA copy number (absolute quantification) using a standard range performed with known quantities of complementary DNA, copies of the RNA of interest.

SECONDARY OUTCOMES:
mRNA expression of caspase-1 | Randomization, 6 and 9 months +/- 8 days post randomisation
  The inflammasome NLRP3 is a multi-protein platform (NLRP3, ASC, pro caspase-1) with an active assembly of inflammatory caspases (notably caspase-1) that cleaves the pro-interleukins IL-1β and IL-18 into mature pro-inflammatory cytokines.
  The biological evaluation criteria will be the mRNA expression of caspase-1 gene in monocytes isolated from peripheral blood measured in cDNA copy number.
mRNA expression of AUC | Randomization, 6 and 9 months +/- 8 days post randomisation
  The inflammasome NLRP3 is a multi-protein platform (NLRP3, ASC, pro caspase-1) with an active assembly of inflammatory caspases (notably caspase-1) that cleaves the pro-interleukins IL-1β and IL-18 into mature pro-inflammatory cytokines.
  The biological evaluation criteria will be the mRNA expression of AUC (apoptotic speck protein containing a caspase recruitment domain) gene in monocytes isolated from peripheral blood measured in cDNA copy number.
mRNA expression of IL-1β | Randomization, 6 and 9 months +/- 8 days post randomisation
  The inflammasome NLRP3 is a multi-protein platform (NLRP3, ASC, pro caspase-1) with an active assembly of inflammatory caspases (notably caspase-1) that cleaves the pro-interleukins IL-1β and IL-18 into mature pro-inflammatory cytokines.
  The biological evaluation criteria will be the mRNA expression of IL-1β in monocytes isolated from peripheral blood measured in copy number.
mRNA expression of IL18 | Randomization, 6 and 9 months +/- 8 days post randomisation
  The inflammasome NLRP3 is a multi-protein platform (NLRP3, ASC, pro caspase-1) with an active assembly of inflammatory caspases (notably caspase-1) that cleaves the pro-interleukins IL-1β and IL-18 into mature pro-inflammatory cytokines.
  The biological evaluation criteria will be the mRNA expression of IL18 in monocytes isolated from peripheral blood measured in copy number.
Plasma level of the pro-inflammatory cytokines IL-1β | Randomization, 6 and 9 months +/- 8 days post randomisation
  The inflammasome NLRP3 is a multi-protein platform (NLRP3, ASC, pro caspase-1) with an active assembly of inflammatory caspases (notably caspase-1) that cleaves the pro-interleukins IL-1β and IL-18 into mature pro-inflammatory cytokines.
  The biological evaluation criteria will be the plasma level of the pro-inflammatory cytokines IL-1β measured by ELISA kits in pg/mL.
Plasma level of the pro-inflammatory cytokines IL18 | Randomization, 6 and 9 months +/- 8 days post randomisation
  The inflammasome NLRP3 is a multi-protein platform (NLRP3, ASC, pro caspase-1) with an active assembly of inflammatory caspases (notably caspase-1) that cleaves the pro-interleukins IL-1β and IL-18 into mature pro-inflammatory cytokines.
  The biological evaluation criteria will be the plasma level of the pro-inflammatory cytokines IL18 measured by ELISA kits in pg/mL.
Plasma level of ultra-sensitive C-reactive Protein | Randomization, 6 and 9 months +/- 8 days post randomisation
  The biological evaluation criteria will be the plasma level of ultra-sensitive C-reactive Protein measured in mg/mL.
Weight loss assessment | Randomization, 6 and 9 months +/- 8 days post randomisation
  Weight measurement in kg
Body mass index assessment | Randomization, 6 and 9 months +/- 8 days post randomisation
  Body mass index measurement
Abdominal perimeter assessment | Randomization, 6 and 9 months +/- 8 days post randomisation
  Abdominal perimeter measurement in centimeters
Hip circumference assessment | Randomization, 6 and 9 months +/- 8 days post randomisation
  Hip circumference measurement in in centimeters
Body composition assessment | Randomization, 6 and 9 months +/- 8 days post randomisation
  Body composition by impedance meter (%)

CONTACTS AND LOCATIONS:
Overall Officials: Rémi NEVIERE, MD, PhD, Study Director — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah M, Hurt RT, Mundi MS. Phenotypes of Obesity: How it Impacts Management. Curr Gastroenterol Rep. 2017 Sep 25;19(11):55. doi: 10.1007/s11894-017-0598-1. PMID 28948512
- [Result] Gruzdeva O, Borodkina D, Uchasova E, Dyleva Y, Barbarash O. Localization of fat depots and cardiovascular risk. Lipids Health Dis. 2018 Sep 15;17(1):218. doi: 10.1186/s12944-018-0856-8. PMID 30219068
- [Result] Pavillard LE, Marin-Aguilar F, Bullon P, Cordero MD. Cardiovascular diseases, NLRP3 inflammasome, and western dietary patterns. Pharmacol Res. 2018 May;131:44-50. doi: 10.1016/j.phrs.2018.03.018. Epub 2018 Mar 26. PMID 29588192
- [Result] Rheinheimer J, de Souza BM, Cardoso NS, Bauer AC, Crispim D. Current role of the NLRP3 inflammasome on obesity and insulin resistance: A systematic review. Metabolism. 2017 Sep;74:1-9. doi: 10.1016/j.metabol.2017.06.002. Epub 2017 Jun 11. PMID 28764843
- [Result] Farhat G, Drummond S, Al-Dujaili EAS. Polyphenols and Their Role in Obesity Management: A Systematic Review of Randomized Clinical Trials. Phytother Res. 2017 Jul;31(7):1005-1018. doi: 10.1002/ptr.5830. Epub 2017 May 11. PMID 28493374
- See also: Obesity and Overweight. WHO 2018 — http://www.who.int/fr/news-room/fact-sheets/detail/obesity-and-overweight
- See also: Thematic files/Environment and health/Esteban — http://invs.santepubliquefrance.fr/Dossiers-thematiques/Environnement-et-sante/Esteban
- See also: Overweight and abdominal obesity in Guadeloupe in 2013 - KANNARI survey — https://ireps.gp.fnes.fr/documentation/consulter-les-ressources-en-ligne-veille/surcharge-ponderale-et-obesite-abdominale-en-guadeloupe-en-2013--kannari-sante-nutrition-et-exposition-au-chlordecone-aux-antilles